CLINICAL TRIAL: NCT04612244
Title: A Prospective Randomized Pivotal Trial of the FARAPULSE Pulsed Field Ablation System Compared With Standard of Care Ablation in Patients With Paroxysmal Atrial Fibrillation
Brief Title: The FARAPULSE ADVENT PIVOTAL Trial PFA System vs SOC Ablation for Paroxysmal Atrial Fibrillation
Acronym: ADVENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CS0934
Record Dates: First submitted 2020-10-26; First posted 2020-11-02 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- FARAPULSE Pulsed Field Ablation System (Experimental)
  Interventions: Device: FARAPULSE Pulsed Field Ablation System
- Force Sensing Radiofrequency Ablation and Cryoballoon Ablation (Active Comparator)
  Interventions: Device: RadioFrequency and Cryoballoon Ablation

INTERVENTIONS:
Device: FARAPULSE Pulsed Field Ablation System — Ablation using the FARAPULSE Pulsed Field Ablation System
  Arms: FARAPULSE Pulsed Field Ablation System
Device: RadioFrequency and Cryoballoon Ablation — Contact Force Enabled RF and Cryoballoon ablation catheters indicated for Paroxysmal Atrial Fibrillation
  Arms: Force Sensing Radiofrequency Ablation and Cryoballoon Ablation

SUMMARY:
This is a prospective, adaptive, multi-center, randomized safety and effectiveness pivotal study comparing the FARAPULSE Pulsed Field Ablation System with standard of care ablation with force-sensing RF catheters and cryoballoon catheters indicated for the treatment of PAF.

ELIGIBILITY:
Key inclusion criteria: Patients are required to meet all the following inclusion criteria to participate in this study:

1. Patients with drug-resistant symptomatic PAF meeting all the following criteria:

   a. Paroxysmal: AF that terminates spontaneously or with intervention within 7 days of onset.

   b. Frequency: i. Physician documentation of recurrent PAF (two or more episodes) within 6 months, AND

   ii. At least one (1) documented episode by a recording such as ECG, EM, Holter monitor or telemetry strip within 12 months of enrollment.

   c. Drug failed: Failed AAD treatment, meaning therapeutic failure of at least one (1) AAD (Class I to IV) for efficacy and / or intolerance.
2. Patients who are ≥ 18 and ≤ 75 years of age on the day of enrollment.
3. Patient who are willing and capable of:

   1. Providing informed consent to undergo study procedures AND
   2. Participating in all examinations and follow-up visits and tests associated with this clinical study.

      Key exclusion criteria:

      Patients will be excluded from participating in this study if they meet any one of the following exclusion criteria:
      * 1. AF that is any of the following:

   <!-- -->

   1. Persistent (both early and longstanding) by diagnosis or continuous duration > 7 days
   2. Requires four (4) or more direct-current cardioversions in the preceding 12 months
   3. Secondary to electrolyte imbalance, thyroid disease, alcohol or other reversible / non-cardiac causes

2. Any of the following atrial conditions:

1. Left atrial anteroposterior diameter ≥ 5.5 cm (by MRI, CT or TTE)
2. Any prior atrial endocardial or epicardial ablation procedure, other than right sided cavotricuspid isthmus ablation or for right sided SVT
3. Any prior atrial surgery
4. Intra-atrial septal patch or interatrial shunt
5. Atrial myxoma
6. Current LA thrombus
7. LA appendage closure, device or occlusion, past or anticipated
8. Any PV abnormality, stenosis or stenting (common and middle PVs are admissible)

   3. At any time, one (1) or more of the following cardiovascular procedures, implants or conditions:

a. Sustained ventricular tachycardia or any ventricular fibrillation

b. Hemodynamically significant valvular disease:

i. Valvular disease that is symptomatic

ii. Valvular disease causing or exacerbating congestive heart failure

iii. Aortic stenosis: if already characterized, valve area < 1.5cm or gradient > 20 mm Hg

iv. Mitral stenosis: if already characterized, valve area < 1.5cm or gradient > 5 mm Hg

v. Aortic or mitral regurgitation associated with abnormal LV function or hemodynamic measurements

c. Hypertrophic cardiomyopathy

d. Any prosthetic heart valve, ring or repair including balloon aortic valvuloplasty

e. Pacemaker, implantable cardioverter defibrillator or cardiac resynchronization therapy devices

f. Any inferior vena cava (IVC) filter, known inability to obtain vascular access or other contraindication to femoral access

g. History of rheumatic fever

h. History of congenital heart disease with any residual anatomic or conduction abnormality

4. Any of the following procedures, implants or conditions:

1. At baseline:

i. New York Heart Association (NYHA) Class III/IV

ii. Left ventricular ejection fraction (LVEF) < 40%

iii. Symptomatic hypotension

iv. Uncontrolled hypertension (SBP > 160 mmHg or DBP > 95 mmHg on two BP measurements at baseline assessment)

v. Symptomatic resting bradycardia

vi. Implantable loop recorder or insertable cardiac monitor,

b. Within the 3 months preceding the Consent Date:

i. Myocardial infarction

ii. Unstable angina

iii. Percutaneous coronary intervention

iv. Heart failure hospitalization

v. Treatment with amiodarone

vi. Pericarditis or symptomatic pericardial effusion

vii. Gastrointestinal bleeding

c. Within the 6 months preceding the Consent Date:

i. Heart surgery

ii. Stroke, TIA or intracranial bleeding

iii. Any thromboembolic event

iv. Carotid stenting or endarterectomy

5. Diagnosed disorder of blood clotting or bleeding diathesis

6. Contraindication to, or unwillingness to use, systemic anticoagulation

7. Patient who is not on anticoagulation therapy for at least 3 weeks prior to the ablation procedure

8. Contraindication to both CT and MRI

9. Sensitivity to contrast media not controllable by premedication

10. Women of childbearing potential who are pregnant, lactating, not using medical birth control or who are planning to become pregnant during the anticipated study period

11. Medical conditions that would prevent participation in the study, interfere with assessment or therapy, significantly raise the risk of study participation, or modify outcome data or its interpretation, including but not limited to:

1. Body Mass Index (BMI) > 40.0
2. Solid organ or hematologic transplant, or currently being evaluated for an organ transplant
3. Severe lung disease, pulmonary hypertension, or any lung disease involving abnormal blood gases or requiring supplemental oxygen
4. Renal insufficiency with an estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2, or any history of renal dialysis or renal transplant
5. Active malignancy or history of treated malignancy within 24 months of enrollment (other than cutaneous basal cell or squamous cell carcinoma)
6. Clinically significant gastrointestinal problems involving the esophagus or stomach including severe or erosive esophagitis, uncontrolled gastric reflux, gastroparesis, esophageal candidiasis or active gastroduodenal ulceration
7. Active systemic infection
8. COVID-19 disease
9. Current confirmed, active COVID-19 disease

ii. Current positive test for SARS-CoV-2

iii. Confirmed COVID-19 disease not clinically resolved at least 3 months prior to the Consent Date.

i. Other uncontrolled medical conditions that may modify device effect or increase risk, including uncontrolled diabetes mellitus (HgbA1c > 8.0% if test result already obtained) or active alcohol abuse

j. Sleep apnea and:

i. An apnea-hypopnea index (AHI) ≥ 15, or

ii. An AHI of ≥ 5 and ≤14 with documented symptoms of excessive daytime sleepiness, impaired cognition, mood disorders or insomnia, or documented hypertension, ischemic heart disease or history of stroke, unless compliant with continuous positive airway pressure (CPAP) treatment.

k. Predicted life expectancy less than one (1) year

12. Clinically significant psychological condition that in the Investigator's opinion would prohibit the subject's ability to meet the protocol requirements

13. Current or anticipated enrollment in any other randomized, interventional or Food and Drug Administration (FDA)-regulated clinical study (data collection for registries or retrospective studies is permitted)

14. Employees / family members of:

1. FARAPULSE or any of its affiliates or contractors
2. The Investigator, sub-Investigators, or their medical office or practice, or healthcare organizations at which study procedures may be performed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Mt. Sinai
Locations (34):
- United States (34):
  - Grandview Medical Center, Birmingham, Alabama
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Banner University Medical Center, Phoenix, Arizona
  - HonorHealth Scottsdale Shea, Scottsdale, Arizona
  - Scripps Memorial Hospital La Jolla, La Jolla, California
  - California Pacific Medical Center, San Francisco, California
  - University of California San Francisco (UCSF), San Francisco, California
  - Emory University Hospital, Atlanta, Georgia
  - St Luke's Regional Medical Center, Boise, Idaho
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital (MGH), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Nebraska Methodist Health system, Inc, Omaha, Nebraska
  - Catholic Medical Center, Manchester, New Hampshire
  - Hackensack University Medical Center/Hackensack Meridian Health, Hackensack, New Jersey
  - NYU Langone Health_Heart Rhythm Center, New York, New York
  - Mount Sinai, Icahn School of Medicine, New York, New York
  - Northwell Health- Lenox Hill Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Providence St Vincent Medical Center, Heart and Vascular Clinical Trials, Portland, Oregon
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - UPMC Pinnacle Health Cardiovascular Institute Inc., Wormleysburg, Pennsylvania
  - Trident Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Saint Thomas Heart at Baptist Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - St Davids_Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - MedStar Washington Hospital Center, Northwest, Washington
  - Swedish Medical Center Heart & Vascular Research, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reddy VY, Mansour M, Calkins H, d'Avila A, Chinitz L, Woods C, Gupta SK, Kim J, Eldadah ZA, Pickett RA, Winterfield J, Su WW, Waks JW, Schneider CW, Richards E, Albrecht EM, Sutton BS, Gerstenfeld EP; ADVENT Investigators. Pulsed Field vs Conventional Thermal Ablation for Paroxysmal Atrial Fibrillation: Recurrent Atrial Arrhythmia Burden. J Am Coll Cardiol. 2024 Jul 2;84(1):61-74. doi: 10.1016/j.jacc.2024.05.001. Epub 2024 May 18. PMID 38864538
- [Derived] Reddy VY, Gerstenfeld EP, Natale A, Whang W, Cuoco FA, Patel C, Mountantonakis SE, Gibson DN, Harding JD, Ellis CR, Ellenbogen KA, DeLurgio DB, Osorio J, Achyutha AB, Schneider CW, Mugglin AS, Albrecht EM, Stein KM, Lehmann JW, Mansour M; ADVENT Investigators. Pulsed Field or Conventional Thermal Ablation for Paroxysmal Atrial Fibrillation. N Engl J Med. 2023 Nov 2;389(18):1660-1671. doi: 10.1056/NEJMoa2307291. Epub 2023 Aug 27. PMID 37634148
- See also: Publication of ADVENT results (PubMed) — https://pubmed.ncbi.nlm.nih.gov/37634148/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 80 Roll-in subjects and 19 randomized subjects (ITT) that withdrew before the procedure.
Units Other Than Participants: procedures
Period: Overall Study
Arm/Group | FARAPULSE Pulsed Field Ablation System | Force Sensing Radiofrequency Ablation and Cryoballoon Ablation
Started | 305; 305 procedures | 302; 302 procedures
Completed | 293; 293 procedures | 290; 290 procedures
Not Completed | 12; 12 procedures | 12; 12 procedures

BASELINE CHARACTERISTICS:
Population: Modified Intention to Treat Subjects with Roll-In subjects and 19 ITT subjects withdrawn prior to the procedure
Groups:
- Total: Total of all reporting groups
Arm/Group | FARAPULSE Pulsed Field Ablation System | Force Sensing Radiofrequency Ablation and Cryoballoon Ablation | Total
Number analyzed (Participants) | 305 | 302 | 607
Age, Continuous [Mean (Full Range); unit: years] | 62.4 [36 to 75] | 62.5 [30 to 75] | 62.4 [30 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 107 | 210
  Male | 202 | 195 | 397
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 11
  Not Hispanic or Latino | 297 | 299 | 596
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 6 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 4 | 11 | 15
  White | 286 | 272 | 558
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 11 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 305 | 302 | 607

OUTCOME MEASURES:

1. Primary Outcome: Composite Safety Endpoint;Proportion of MITT Subjects With One or More of the Specified Device or Procedure Related SAEs
Description: Proportion of Intent to Treat subjects with one or more of the specified device or procedure related SAEs
Time Frame: 7 days and 12 Months
Population: MITT
Measure: Count of Participants; unit: Participants
Arm/Group | FARAPULSE Pulsed Field Ablation System | Force Sensing Radiofrequency Ablation and Cryoballoon Ablation
Number analyzed (Participants) | 305 | 302
Participants | 6 | 4

2. Primary Outcome: Primary Effectiveness Endpoint
Description: Treatment Success: The primary effectiveness endpoint is Treatment Success in MITT Subjects, defined as:
  1. Acute Procedural Success AND
  2. Chronic Success, defined as freedom from:
     1. At the Index / Rescheduled Index Procedure: Use of a non-randomized treatment modality for PVI
     2. After the Blanking Period:
     i. Occurrence of any Detectable AF, AFL or AT (excluding CTI-dependent flutter confirmed by EP study)
     ii. Any cardioversion for AF, AFL or AT (excluding for CTI-dependent flutter)
     iii. Use of any Type I or Type III antiarrhythmic medication for the treatment of AF, AFL or AT
     c. At any time:
     i. Re-ablation for AF, AFL or AT (other than for CTI-dependent flutter)
     ii. Use of amiodarone, except intra-procedurally to control an arrhythmia Endpoint status will be assessed through the Month 12 Assessment (Day 360 ± 30).
Time Frame: 12-Months
Population: MITT
Measure: Count of Participants; unit: Participants
Arm/Group | FARAPULSE Pulsed Field Ablation System | Force Sensing Radiofrequency Ablation and Cryoballoon Ablation
Number analyzed (Participants) | 305 | 302
Participants | 204 | 194
Statistical Analysis 1: Comparison: FARAPULSE Pulsed Field Ablation System vs Force Sensing Radiofrequency Ablation and Cryoballoon Ablation; The primary effectiveness endpoint for this study is Treatment Success, which will be analyzed as a test of non-inferiority of the event rate at 12 months using a noninferiority margin of 15%. The null and alternative hypotheses are: H0: PT ≤ PC - 0.15 versus HA: PT > PC - 0.15 where PT is the Treatment Success rate at 12 months in the Pulsed Field Group and PC is the Treatment Success rate at 12 months in the Thermal (Control) Group; Test type: Non-Inferiority — PT will be deemed to be non-inferior to PC if it can be established that the posterior probability Pr(HA | data) > Ψeff, where Ψeff is a pre-specified threshold value that controls the one-sided type I error rate (under simulation) at level 0.05. In the absence of missing data, the posterior distributions for PT and PC would be conjugate Beta distributions; p = 0.05, t-test, 1 sided

3. Secondary Outcome: Change in PV Cross-sectional Area
Description: Mean change in aggregate PV Cross-Sectional area (cm^2) from baseline to Day 90
Time Frame: 3 months
Population: MITT
Measure: Mean (95% Confidence Interval); unit: cm^2.
Arm/Group | FARAPULSE Pulsed Field Ablation System | Force Sensing Radiofrequency Ablation and Cryoballoon Ablation
Number analyzed (Participants) | 259 | 255
cm^2. | -0.18 [-0.37 to 0.00] | -1.18 [-1.39 to -0.97]

4. Secondary Outcome: Primary Effectiveness Treatment Success Tested for Superiority
Description: The secondary effectiveness endpoint is the same as the primary effectiveness endpoint but will be tested for superiority rather than non-inferiority. The proportion of Pulsed Field Subjects with Treatment Success will be assessed for superiority to the proportion of Thermal Subjects with Treatment Success.
Time Frame: 12 Months
Population: MITT
Measure: Number (95% Confidence Interval); unit: Treatment Success Rate
Arm/Group | FARAPULSE Pulsed Field Ablation System | Force Sensing Radiofrequency Ablation and Cryoballoon Ablation
Number analyzed (Participants) | 305 | 302
Treatment Success Rate | 73.3 [68.1 to 78.1] | 71.3 [66.0 to 76.3]
Statistical Analysis 1: Comparison: FARAPULSE Pulsed Field Ablation System vs Force Sensing Radiofrequency Ablation and Cryoballoon Ablation; The secondary effectiveness endpoint for the ADVENT Trial is Treatment Superiority uses the same definition as the primary effectiveness endpoint for Treatment Success, but the test is for superiority between MITT subjects in the PFA and Thermal Groups; Test type: Superiority — The null and alternative hypotheses are provided below. H0: PT ≤ PC versus HA: PT > PC where PT is the Treatment Success rate at 12 months in the Pulsed Field Group, and PC is the Treatment Success rate at 12 months in the Thermal Group. Modeling will be identical primary endpoint and superiority concluded if the posterior probability Pr(HA | data) > Ψeff, sup, where the threshold Ψeff,sup is a pre-specified threshold value that controls the one-sided type I error rate at level 0.025; p = 0.025, t-test, 1 sided; Median Difference (Final Values) = 0.708

ADVERSE EVENTS:
Time Frame: 420 days
Arm/Group | FARAPULSE Pulsed Field Ablation System | Force Sensing Radiofrequency Ablation and Cryoballoon Ablation
All-Cause Mortality (participants affected / at risk) | 2/305 | 1/302
Serious Adverse Events (participants affected / at risk) | 37/305 | 34/302
Other Adverse Events (participants affected / at risk) | 88/305 | 103/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FARAPULSE Pulsed Field Ablation System (N=305) | Force Sensing Radiofrequency Ablation and Cryoballoon Ablation (N=302)
Patient Condition-Non Cardiovascular-Other (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Atrial Fibrillation (Cardiac disorders) | 6 (7) | 9 (11)
Atrial Flutter (Cardiac disorders) | 2 (3) | 1 (1)
Atrial Flutter-Not Specified (Cardiac disorders) | 1 (1) | 1 (1)
Atrial Tachycardia Other SVT (Cardiac disorders) | 0 (0) | 1 (1)
Atypical (Type II) Atrial Flutter (Cardiac disorders) | 1 (2) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Tamponade- Unrelated to Procedure/Device (Cardiac disorders) | 0 (0) | 1 (1)
Chest Pain Other (Cardiac disorders) | 1 (1) | 0 (0)
Conduction Disturbances/ Arrhythmia-Other (Cardiac disorders) | 1 (2) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0)
Left Atrial (Type II, Atypical) Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Perforation with Tamponade (Cardiac disorders) | 2 (2) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
SinuasBradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Symptomatic Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0)
Intracardiac Thrombus (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
HEENT (Eye disorders) | 1 (1) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 2 (2) | 2 (2)
Hemorrhage Unrelated to Procedure (Gastrointestinal disorders) | 0 (0) | 1 (1)
EP/ ablation Other- Multi Organ Failure (General disorders) | 1 (1) | 0 (0)
Pain Cardiovascular (Non-Ischemic) (General disorders) | 0 (0) | 1 (1)
Hemorrhage Unelated to Procedure (General disorders) | 0 (0) | 1 (1)
Pericarditis (General disorders) | 1 (1) | 0 (0)
Gastrointestinal (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cancer (Infections and infestations) | 1 (1) | 0 (0)
Coronavirus Infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal (Infections and infestations) | 2 (2) | 1 (1)
Localized Infection (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Systemic Infection (Infections and infestations) | 2 (2) | 1 (1)
Access Site Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Musculoskeletal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Oozing/Bleeding (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Physical Trauma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Procedure Related Hypertension (Investigations) | 1 (1) | 0 (0)
Abnormal Lab Values (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pulmonary Edema (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Whole Body Other (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Gastrointestinal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral Vascular Accident (Nervous system disorders) | 0 (0) | 1 (1)
Neurological (Nervous system disorders) | 0 (0) | 2 (2)
Syncope (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transient Ischemic Attack (Nervous system disorders) | 1 (1) | 1 (1)
Psychological (Psychiatric disorders) | 0 (0) | 1 (1)
Procedure Related Genitourinary (Renal and urinary disorders) | 1 (1) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Integumentary (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Vascular disorders) | 0 (0) | 1 (1)
Death (Vascular disorders) | 0 (0) | 1 (1)
Fistula (Arterial/Venous) (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FARAPULSE Pulsed Field Ablation System (N=305) | Force Sensing Radiofrequency Ablation and Cryoballoon Ablation (N=302)
Atrial Fibrillation (Cardiac disorders) | 12 (15) | 22 (27)
Gastrointestinal (Gastrointestinal disorders) | 12 (13) | 15 (18)
Coronavirus infection (Infections and infestations) | 30 (30) | 37 (37)
Post Procedure Wound Discomfort (Injury, poisoning and procedural complications) | 19 (19) | 8 (8)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 15 (16) | 21 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT04612244/Prot_002.pdf
  • Statistical Analysis Plan (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/44/NCT04612244/SAP_001.pdf